CLINICAL TRIAL: NCT03391219
Title: Combined Intravitreal Injection of Bevacizumab and Fasudil Versus Bevacizumab Alone for Macular Edema Secondary to Retinal Vein Occlusion in Previously Treated Patients.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96299
Record Dates: First submitted 2017-12-19; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravitreal Bevacizumab (Active Comparator)
  Interventions: Drug: injection bevacizumab
- intravitreal Bavacizumab and Fasudil (Active Comparator)
  Interventions: Drug: injection Combined Bevacizumab and Fasudil

INTERVENTIONS:
Drug: injection bevacizumab — 1.25 mg/0.05 cc bevacizumab
  Arms: intravitreal Bevacizumab
Drug: injection Combined Bevacizumab and Fasudil — 1.25 mg/0.05 cc bevacizumab and 0.15mg/0.05 cc fasudil
  Arms: intravitreal Bavacizumab and Fasudil

SUMMARY:
This study is aimed to compare the effect of combined intravitreal Bevacizumab and Fasudil injection with Bevacizumab only injection in patients with persistant macular edema secondary to ratinal vein occlusion.

Methods:

In this study patients with retinal vein occlusion patient who had at least three or more intravitreal AntiVEGF injection with persistence of macular edema at funduscopic examination is recruited. The eligible patients in randomized in two groups "Bevacizumab" and "Bavacizumab + Fasudil" and in injected intravitreally for 3 times monthly. In "Bevacizumab+Fasudil" group patients receive two injections at each session Bavacizumab and Fasudil. In "Bevacizumab" group patients receive only Bevacizumab. The patients are followed for 6 months and central macular thickness and visual acuity is measured at baseline and monthly for 6 month. Baseline ancillary exams include Fluorescein Angiography and OCT-Angiography which is performed at the final exam as well. Patients needing any therapeutic intervention is addressed during the 6 month follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Branch retinal vein or central retinal vein occlusion Previous at least 3 intravitreal antiVEGF injection Macular edema in SD-OCT CMT = >250 microns BCVA equal or lesd than 20/40

Exclusion Criteria:

* Moderate or severe corneal opacity Significant cataract obscuring retinal exam or OCT Glaucoma History of vitreoretinal surgery Diabetic retinopathy Macular disease (AMD,ERM,VMT Kidney or Liver disease Uncontrolled or moderate or severe Anemia Uncontrolled hypertention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Measure Macular Thickness | 9 month
  Optical Coherence Tomography

SECONDARY OUTCOMES:
Measure Visual acuity | 9 month
  Snellen chart

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran